CLINICAL TRIAL: NCT00970736
Title: Corticobulbar Motor Output in Aging Adults
Brief Title: Stability of Motor Output in Aging Adults
Status: Completed | Type: Observational
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Other Study IDs: C6697-M
Record Dates: First submitted 2009-09-01; First posted 2009-09-02 (Estimated); Results first posted 2015-04-08 (Estimated); Last update posted 2015-04-08 (Estimated); Status verified 2014-12

CONDITIONS: Swallowing
Keywords: Motor cortex; Motor control; Neuroplasticity; Aging; Swallowing

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: 20 healthy participants between 60 and 80 years of age. Ten men and 10 women.

SUMMARY:
The goal of this project is to examine the area of the brain that controls muscle movement for a group of muscles important for swallowing, and to see how that area changes over 2 weeks of time.

DETAILED DESCRIPTION:
A large number of our nation's veterans develop dysphagia due to the myriad of potential etiological sources of swallowing disorders, including stroke and head and neck cancer. The Veteran's Health Administration has recently identified dysphagia as a major clinical focus for the VA system (Sullivan & Dennis, 2006). In order to accurately assess adaptations in motor cortex, it is first necessary to have a reliable tool for measuring organizational representation in the motor cortex. Transcranial magnetic stimulation (TMS) is a desirable choice for such measurement because of the ability to identify causative relationships between an area of motor cortex stimulated and muscle response. Therefore, the specific research objectives of this proposal are:

1. To demonstrate the reproducibility of TMS mapping of the submental muscle group in healthy older adults between 60 and 80 years of age
2. To determine the neural representation of submental musculature in the motor cortex of healthy older adults between 60 and 80 years of age.

Twenty healthy adults, 10 men and 10 women, between the ages of 60 and 80 years will serve as research participants. TMS will be used to establish motor maps of the submental muscles. Subjects will undergo two testing sessions, on day 1 and day 14. The results from each session will be compared to assess excitability and representation within the motor cortex, and to assess stability and reliability of measurement.

ELIGIBILITY:
Inclusion Criteria:

* Between 60 and 80 years of age

Exclusion Criteria:

* History of dysphagia
* History of neurologic disease
* History of head or neck cancer
* History of stroke
* Untreated hypertension
* History of a heart condition or heart disease
* Currently pregnant
* Contraindication to TMS including:

  * Metallic hardware on the scalp in the area where TMS will be applied
  * Cardiac pacemaker
  * Implanted medication pumps or an intracardiac line
  * Prior diagnosis of seizure or epilepsy in the subject (childhood history of benign febrile seizure will not be a contraindication)
  * Poorly controlled migraine headaches
  * Previous brain neurosurgery
  * Medications that can lower seizure threshold (Appendix B)
  * Unstable medical conditions
  * Lowest motor thresholds above 80% on TMS

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy adults between 60 and 80 years of age
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2009-11; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Karen Hegland, PhD, Principal Investigator — North Florida/South Georgia Veterans Health System
Locations (1):
- North Florida/South Georgia Veterans Health System, Gainesville, Florida, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Healthy Participants: 20 healthy participants between 60 and 80 years of age. Ten men and 10 women.
Period: Overall Study
Arm/Group | Healthy Participants
Started | 20
Completed | 18
Not Completed | 2

BASELINE CHARACTERISTICS:
Population: Healthy adults between the ages of 60 and 80 years
Arm/Group | Healthy Participants
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 4
  >=65 years | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 68 (6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 10
Region of Enrollment [Number; unit: participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: Mean Motor Evoked Potential Amplitude for Submental Cortical Representation
Description: Cortical sites are stimulated sequentially from the SOLMT in the anterior direction. At each site, 5 pulses of 110% of the MEP threshold obtained at the SOLMT are delivered and recorded. If a site produces no MEP in 3/5 pulses it is considered non-submental. This process is continued until the entire submental representation is surrounded by non-submental responsive sites. The number of sites is used to calculate the area of submental representation. The mean sEMG amplitudes of the submental muscles for each of these sites is then calculated for the mean MEP measure.
Time Frame: 2 weeks
Population: This data was not analyzed because the study funding, as well as PIs VA affiliation, ended prior to any data analyses.
Arm/Group | Healthy Participants
Number analyzed (Participants) | 0

2. Secondary Outcome: Motor Map Center of Gravity
Description: Position on the TMS motor map with highest amplitude response to stimulation in the muscles of interest (submental muscles).
Time Frame: 2 weeks
Population: This data was not analyzed because the study and funding, as well as the PIs VA affiliation, ended prior to doing any analyses.
Arm/Group | Healthy Participants
Number analyzed (Participants) | 0

3. Secondary Outcome: Area of Submental Representation
Description: Cortical sites are stimulated sequentially from the SOLMT in the anterior direction. At each site, 5 pulses of 110% of the MEP threshold obtained at the SOLMT are delivered and recorded. If a site produces no MEP in 3/5 pulses it is considered non-submental. This process is continued until the entire submental representation is surrounded by non-submental responsive sites. The number of sites is used to calculate the area of submental representation.
Time Frame: 2 weeks
Population: This data was not analyzed because the study, funding, and PIs VA affiliation ended prior to any data analyses.
Arm/Group | Healthy Participants
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 2 weeks (time including the day 1 testing, day 2 testing, and time in between).
Arm/Group | Healthy Participants
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No